CLINICAL TRIAL: NCT06174389
Title: Physiological Changes Underlying the Weight Loss Plateau in Human
Brief Title: ADAPT Study: Assessing Diet, Appetite and Physiology Throughout Weight Loss Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ellen Schur, MD, MS, Professor: School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00017667; R01DK134417 (NIH)
Record Dates: First submitted 2023-11-13; First posted 2023-12-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: Gloisis; Weight Change
MeSH Terms: conditions — Obesity; Body Weight Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral Weight Loss (Experimental): Participants will undergo a behavioral weight loss program.
  Interventions: Behavioral: Behavioral Weight Loss Program

INTERVENTIONS:
Behavioral: Behavioral Weight Loss Program — Behavioral Weight Loss Program is a modified version of the Diabetes Prevention Program.

SUMMARY:
Behavioral weight loss programs for obesity can result in weight loss and health benefits. However, behavioral weight loss often stops despite efforts to continue losing weight, this can be called an involuntarily weight loss plateau. This study investigates changes in metabolism and/or the brain that contribute to the occurrence of an involuntary weight loss plateau.

DETAILED DESCRIPTION:
Participants will be asked to enroll for 18-months. Each participant will complete 3 in-person study visits, then participate an a 6-month weight loss program delivered remotely. Some participants may be invited to complete 3 additional in-person visits. Study Visit activities include questionnaires, blood draws, brain MRIs, body measurement and dual energy x-ray absorptiometry (DXA) scan for body composition measurement, a breathing test, and biopsies of muscle and fat tissue. Each participant will be provided a fitness tracker and body weight scale to use throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30.0 - 50.0 kg/m2
* Able to attend study intervention classes and study visits/assessments
* Independently living with access to food preparation facilities

Exclusion Criteria:

* Current smoker or regular use of nicotine containing products and/or cannabis
* Heavy alcohol use (≥2 drinks/d for females, ≥3 drinks/d for males) or drug use
* Known cognitive impairments or h/o stroke
* Type 2 diabetes (known diagnosis or by screening A1c (≥6.5%))
* Medical conditions (chronic diseases, cancer, MS) or labs limiting ability to participate
* Females: currently pregnant (or 6-months postpartum of full-term pregnancy) and/or current breastfeeding
* Use of medications with significant effects on appetite (e.g., weight loss medications, atypical antipsychotics, stimulants) and/or chronic use of anticoagulants
* History of bariatric surgery
* History of eating disorder
* Current participation in a formal weight loss program
* Prior or current participation in a research study involving weight loss
* Weight-reduced by >10% within past year
* Weight > 330 pounds (MRI limit)
* Allergy or intolerance to or unwillingness to consume study foods provided at visit
* MRI contraindication (e.g., implanted metal, claustrophobia)
* Do not have a phone compatible with activity tracker or access to videoconferencing platform that will be used for the dietary intervention or other appropriate technology needed to complete study procedures
* Any condition(s) found by the study team and confirmed with the PI(s) that make it unsafe to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in maximal respiratory capacity (oxygen consumption rate) in peripheral blood mononuclear cells | From baseline to active weight loss (at least 21 days of weight loss equivalent or greater than 0.5 pounds per week) and from baseline to weight loss plateau (after active weight loss, at least 21 days of halted weight loss, or +/- 0.25 pounds/week).
  Mitochondrial maximal respiratory capacity will be measured in fasting samples from peripheral blood mononuclear cells.
Change in fMRI BOLD signal | From baseline to a weight loss plateau (after active weight loss, at least 21 days of halted weight loss, or +/- 0.25 pounds/week).
  fMRI BOLD signal to visual food cues within a priori brain regions of interest pre and post consuming a standardized meal. Meal-induced change will be calculated by post-pre meal BOLD signal.
Entry into involuntary weight loss plateau | throughout 18-month enrollment
  binary outcome (Y/N) and time from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Schur, MD, MS, Principal Investigator — University of Washington; Marian Neuhouser, PhD, RD, Principal Investigator — Fred Hutch Cancer Center
Locations (2):
- United States (2):
  - Fred Hutch Cancer Center, Seattle, Washington
  - University of Washington - South Lake Union, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No